CLINICAL TRIAL: NCT06421779
Title: A Game-Like Skin Testing Experience: The Effect of Virtual Reality (VR) on Skin Prick Test Related Pain and Fear in Children (Randomized Controlled Trial)
Brief Title: The Effect of Virtual Reality (VR) on Skin Prick Test Related Pain and Fear in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Cihangir Sahin, Research Assistant Medical Doctor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADUPIA-CSAHIN-1
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Pain; Fear; Fear of Pain; Child, Only; Allergy
Keywords: Skin Prick Test; Virtual Reality; Pain; Fear; Child; Allergy
MeSH Terms: conditions — Pain; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: A Prospective parallel group randomized controlled trial.
Who Masked: Participant
Masking Description: Children aged 4 to 10 years for whom a skin prick test has been decided.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VR (Experimental): Children in the VR group put on VR glasses for approximately two minutes before the skin prick test and watched a VR underwater experience video throughout the procedure.
  Interventions: Behavioral: Virtual reality (VR)
- No Intervention: Control (No Intervention): Children in the control group underwent a routine skin prick test procedure. Control group children did not receive any distraction techniques.

INTERVENTIONS:
Behavioral: Virtual reality (VR) — Children watch underwater experience video by wearing the virtual reality glass during the skin prick test.
  Arms: Experimental: VR

SUMMARY:
This study aims to show the effect of VR on skin prick test-related pain and fear in children. The investigators will compare the effect of VR on skin prick test-induced pain and fear in children applying to the Pediatric Allergy outpatient clinic with controls who underwent skin prick test without the use of VR.

DETAILED DESCRIPTION:
Pain and fear during interventional procedures in pediatric patients are some of the most difficult problems in hospitals. While bad experiences in childhood can lead to increased sensitivity to pain, sleep problems, social learning difficulties, phobias, pre-treatment anxiety disorders, and treatment resistance; increases the risk of anxiety and depression in adulthood.

Skin prick test is the gold standard diagnostic method most frequently used in Pediatric Allergy clinics for the detection of allergens with high sensitivity, specificity, and reliability. The numerous pricking procedures performed during the skin test may turn into a painful and frightening experience for children.

Virtual reality (VR) is often accomplished using a special headset or glasses and can create for children a virtual world separate from their current physical environment, effectively distracting them from the possible pain and fear experience.

There is no study in the literature investigating the effect of VR on skin prick test-related pain and fear in children. This study aims to show the effect of VR on skin prick test-related pain and fear in children. The investigators will compare the effect of VR on skin prick test-induced pain and fear in children applying to the Pediatric Allergy outpatient clinic with controls who underwent skin prick test without the use of VR.

The hypotheses of this study were to:

H1: The virtual reality (VR) group will experience less pain due to the skin prick test than the control group.

H2: The virtual reality (VR) group will experience less fear due to the skin prick test than the control group.

Study Design:

This study is a parallel group randomized controlled trial planned to be conducted in the skin testing unit of a tertiary reference center of a pediatric allergy outpatient clinic between March and June 2024. The CONSORT guideline will be followed in the study. Fifty children between the ages of 4 and 10 years, who decided to undergo skin prick testing, will be randomized into two groups: using VR (VR group, n = 25) and not using VR (Control group; n = 25) by block randomization method. The reason for choosing this age group is that this age group is the common validation age range of the Wong-Baker FACES Pain Rating Scale (WB-FACES) and Child Fear Scale (CFS), which the investigators will use in the evaluation of pain and fear, in the Turkish children. At the same time, children in this age group are curious about technology and open to collaboration.

Sample Size and Randomization:

The number of patients was determined by taking the data obtained from the reference study titled "The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy® (Randomized Controlled Trial)". Power analysis was performed based on self-report data of the WB-FACES Pain Rating scale in the study. According to the calculation by G*Power 3.1.9.7, the effect size was determined as 0.92, the alpha margin of error was 0.05, the statistical power was 80%, and it was determined that at least 19 participants in each group were required to conduct the study. The analysis showed that a total sample size of 38 participants would be sufficient to detect significant differences. In light of the potential losses of 10% that may occur during the study, the investigators planned to include at least 21 participants in both groups to obtain a total of 42 participants.

In the literature, the studies show that gender and age affect pain and fear associated with invasive procedures in children. Therefore, gender (girls and boys) and age group (4-6 years (preschool) and 7-10 years (school age)) variables were used for block randomization. Blocks were repeated 5 times in each group. 25 participants were assigned to each of the VR and Control groups. A blocked randomization list was developed using an online randomization tool. The investigators were not blinded to group allocation because they performed the randomization themselves.

Ethics:

The study was approved by the local research ethics committee of our institution (2024/66). All participants will take part voluntarily, and personal written informed consent will be obtained from the parents of all participants, and verbal consent will be obtained from the participants before participation.

Data Collection Tools:

Data will be collected with a case report form created using WB-FACES and CFS. Both scales are suitable for personal, parent, and researcher evaluation. In our study, children's personal, parent, and researcher reporting data will be evaluated for both scales. Investigator reporting data will be evaluated by a specialist nurse trained on the scales.

Wong-Baker FACES Pain Rating Scale (WB-FACES):

The Wong-Baker FACES Pain Rating Scale (WB-FACES) was developed in 1981 and revised in 1983. WB-FACES is a reliable scale that has been validated for the Turkish population. The scale is used to diagnose pain in children ages 3-18 years. It consists of six facial expressions, each representing increasing degree of pain scored from 0 to 10 from left to right (0 = very happy face/no pain, 10 = a crying face/worst pain imaginable). High scores indicate low pain tolerance. The child is asked to rate his/her pain by asking "Can you show me the face that shows how you feel right now?".

Children's Fear Scale (CFS):

The Child Fear Scale (CFS) was developed in 2011. It was adapted into Turkish in 2018, by studying it with children aged 4-10 years. It consists of five facial expressions representing a range from neutral=0 to extreme fear=4.

Virtual Reality (VR):

Virtual reality (VR) allows the user to visit a three-dimensional world, isolating them from real life. VR is an advanced technology that offers a 360-degree visual and audio simulation that surrounds the user and allows them to look in all directions. In this study, VR intervention will be performed using a smartphone (Samsung Galaxy S23 Ultra, Qualcomm Snapdragon 8 Gen 2 processor, 12 GB RAM, Android 14 version, One UI 6.0 version, Dynamic AMOLED 1440x3088 QHD+ Pixel Screen, Stereo Dual Speakers), VR glasses (Schulzz VRG Pro) and a VR underwater experience video (2160p resolution video suitable for VR format) that will attract the attention of age groups.

Procedure:

Each child will be admitted to the skin testing unit with his/her parents. The skin testing unit has the same environmental conditions (seat, temperature, light, noise, etc.). Participants will be randomly selected into groups. The researcher will inform the participants and parents about the skin prick test and scales (WB-FACES and CFS). Before the procedure, all participants will be asked verbally about their baseline fear status due to the skin prick test.

Participants in the VR group will put on VR glasses for approximately two minutes before the skin prick test and watch a VR underwater experience video throughout the procedure. Participants in the control group will undergo a routine skin prick test procedure. The VR intervention and skin prick testing will terminate at the same time. The researcher will use a case report form to collect data for participants and their parents. Immediately after the procedure, participants will describe their pain levels with WB-FACES and their fear levels with CFS. Meanwhile, a volunteer parent and a specialist nurse will observe the children's behavior and perform the WB-FACES and CFS evaluations separately. The data collection process will be planned to be completed in approximately ten minutes.

Skin prick test:

Skin prick tests will be performed over the same period by a volunteer nurse with at least 5 years of experience. All participants will undergo the same aeroallergen skin test panel. Skin prick tests will be performed using a prick test applicator (MedBlue One, Türkiye) on the flexural aspect of the forearm by standard guidelines using standardized glycerinated extracts (1% weight/volume) from LOFARMA (Milan, Italy).

Statistical analysis:

SPSS version 23.0 statistical software (IBM SPSS Inc., Chicago, IL, USA) will be used for statistical analysis. Categorical variables will be presented as numbers (%), and continuous variables will be presented as mean±SD and median values (interquartile range-IQR). Univariate analyses including categorical data will be performed using the χ2 test. If data exhibit normality according to the Shapiro-Wilk normality test, parametric values will be analyzed using the Student's t-test, and non-parametric variables will be analyzed using the Mann-Whitney U test. P<0.05 value was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 4-10 years
* requirement of skin prick test due to allergic diseases

Exclusion Criteria:

* having chronic diseases (except allergic diseases)
* vision, hearing, and speech disorders
* psychiatric and neurological diseases
* mental status disorder, learning and perception disorder
* a history of pre-procedure sedative, analgesic or narcotic drug use within 24 hours
* a history of active infection
* those who are scheduled to undergo a skin test other than an aeroallergen panel
* contra-indicated conditions for skin prick testing such as dermographism, severe eczema, being under drugs (immunosuppressive drugs, antihistamine, steroid, etc)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Skin prick test-related pain | Through painful procedure completion, an average of 10 minutes.
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. The Wong-Baker FACES Pain Rating Scale (WB-FACES) was developed in 1981 and revised in 1983. WB-FACES is a reliable scale that has been validated for the Turkish population. The scale is used to diagnose pain in children ages 3-18 years. It consists of six facial expressions, each representing increasing degree of pain scored from 0 to 10 from left to right (0 = very happy face/no pain, 10 = a crying face/worst pain imaginable). High scores indicate low pain tolerance. The child is asked to rate his/her pain by asking "Can you show me the face that shows how you feel right now?".
Skin prick test-related fear | Through fearful procedure completion, an average of 10 minutes.
  The Child Fear Scale (CFS) used. The Child Fear Scale (CFS) was developed in 2011. It was adapted into Turkish in 2018, by studying it with children aged 4-10 years. It consists of five facial expressions representing a range from neutral=0 to extreme fear=4.

CONTACTS AND LOCATIONS:
Overall Officials: Cihangir Sahin, Study Director — Aydin Adnan Menderes University, Department of Pediatric Immunology and Allergy, Aydin, Türkiye
Locations (1):
- Aydin Adnan Menderes University, School of Medicine, Department of Pediatric Immunology and Allergy, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahin C, Cinakli S, Atar Bese S, Tuncerler G, Torer N, Erge D, Uysal P. The effect of virtual reality on skin prick test-related pain and fear in children: a randomized controlled trial. Eur J Pediatr. 2025 Jun 18;184(7):427. doi: 10.1007/s00431-025-06262-x. PMID 40528065